CLINICAL TRIAL: NCT01732328
Title: Calcium Plus Vitamin D Supplementation During Pregnancy of Adolescent Mothers: Effects on Maternal and Infant Bone Mass, Calcium and Bone Metabolism and Breast Milk Composition
Brief Title: Effect of Calcium Plus Vitamin D Supplementation on Adolescent Mother and Infant Bone Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Flavia Fioruci Bezerra, DSc, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE 0002.0361.000-09; CNPq (Other Grant/Funding Number: 471872/08-3)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Lactation Bone Loss; Infant Bone Growth
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Inactive pill (microcrystalline cellulose and corn starch) taken daily
- Calcium plus vitamin D (Active Comparator): 600mg of calcium and 200 international units (IU) vitamin D taken daily
  Interventions: Dietary Supplement: Calcium plus vitamin D

INTERVENTIONS:
Dietary Supplement: Calcium plus vitamin D
  Arms: Calcium plus vitamin D

SUMMARY:
Pregnancy and lactation are periods of high calcium requirement. Inadequate maternal calcium intake and vitamin D insufficiency may adversely affect fetal and neonatal growth and maternal bone mass particularly in adolescent mothers. The investigators propose to evaluate the influence of calcium plus vitamin D supplementation during pregnancy on bone mass of lactating adolescent mothers with habitually low calcium and vitamin D, on fetal growth and neonate bone mass. Mothers are randomly assigned to receive daily calcium (600 mg) plus vitamin D3 (200 IU) supplement or placebo from mid gestation until parturition. Fetal growth parameters are assessed by standard ultrasound techniques at mid and late gestation. Maternal bone mass is assessed by dual energy x-ray absorptiometry (DXA) at 2 and 5 months postpartum and 6 months after weaning. Infant bone mass is assessed by DXA at 2 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 y old
* between 23 and 29 wk of gestation
* primiparous
* carrying single fetus
* intending to exclusively or predominantly breastfeed

Exclusion Criteria:

* chronic health problems
* smokers
* users of nutritional supplements, except iron supplements provided during standard prenatal care

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Differences in maternal bone mass changes postpartum between supplemented and placebo groups | 2, 5 and 12 months postpartum
Differences in fetal growth and infant bone mass between supplemented and placebo groups | 2nd and 3rd trimester gestation and 2 mo postpartum

SECONDARY OUTCOMES:
Differences in changes of bone and calcium related hormones and vitamin D status between supplemented and placebo groups | 2nd and 3rd trimester of pregnancy and 2, 5, 12 mo postpartum
Differences in human breast milk composition (nutrients and hormones) between supplemented and placebo groups | 2 months postpartum
Differences in maternal bone status according to vitamin D receptor (VDR) polymorphisms | 2, 5 and 12 months postpartum
Differences in infant body composition between supplemented and placebo groups | 2 months postpartum
Differences in changes of maternal body composition postpartum between supplemented and placebo groups | 2, 5 and 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Flavia F Bezerra, DSc, Principal Investigator — Universidade do Estado do Rio de Janeiro, Brazil; Carmen M Donangelo, PhD, Study Director — Universidade Federal do Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Rached V, Diogenes MEL, Donangelo CM, Bezerra FF. Calcium plus vitamin D supplementation during pregnancy reduces postpartum fat mass in adolescents: A randomized trial. Am J Hum Biol. 2023 Sep;35(9):e23911. doi: 10.1002/ajhb.23911. Epub 2023 May 11. PMID 37166151
- [Derived] Diogenes ME, Bezerra FF, Rezende EP, Donangelo CM. Calcium Plus Vitamin D Supplementation During the Third Trimester of Pregnancy in Adolescents Accustomed to Low Calcium Diets Does Not Affect Infant Bone Mass at Early Lactation in a Randomized Controlled Trial. J Nutr. 2015 Jul;145(7):1515-23. doi: 10.3945/jn.114.208140. Epub 2015 May 27. PMID 26019245
- [Derived] Diogenes ME, Bezerra FF, Rezende EP, Taveira MF, Pinhal I, Donangelo CM. Effect of calcium plus vitamin D supplementation during pregnancy in Brazilian adolescent mothers: a randomized, placebo-controlled trial. Am J Clin Nutr. 2013 Jul;98(1):82-91. doi: 10.3945/ajcn.112.056275. Epub 2013 May 29. PMID 23719547